CLINICAL TRIAL: NCT04936789
Title: Clinical Feasibility of the IMES Transradial Prosthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP2020072116
Record Dates: First submitted 2021-06-07; First posted 2021-06-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single arm. All subjects will receive the intervention. Comparator device will be subjects' own prosthesis at baseline.
  Interventions: Device: IMES

INTERVENTIONS:
Device: IMES — Surgical implantation of IMES

SUMMARY:
This study will evaluate the feasibility of using implanted myoelectric sensors (IMES) to control a transradial prosthesis

DETAILED DESCRIPTION:
The study assesses the feasibility of an implantable myoelectric prosthesis control system to control a transradial prosthesis. Implantable Myoelectric Sensors (IMES) will be implanted into the residual forearm muscles of three transradial amputee subjects. These devices wirelessly transmit electrical muscle signals to an electromechanical prosthetic wrist and hand.

Following a two-week recovery from implantation of up to 16 IMES into residual forearm muscles, subjects will begin a two week training phase. When they receive their custom-fit IMES Transradial Prosthesis (including electromechanical wrist and hand) subjects initiate approximately four months of home use. Subjects will be offered up to five post-study follow-up visits. The usability and functionality of the prosthetic system will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* (unilateral acquired transradial) amputation
* residual limb size requirements to fit investigational device componentry
* at least 6 residual muscle locations available for implantation
* good compliance with health service (rehabilitation)
* willing to undergo surgical implantation of IMES Sensor implants
* experience with myoelectric upper limb prostheses
* using own myoelectric device approximately 6-8h/day
* able to provide informed consent and attend the study visits

Exclusion Criteria:

* any condition which in the opinion of the investigator poses a risk to health
* neurological disorder that may prohibit accurate control
* major injury proximal to the level of amputation
* neuromuscular disorder
* nerve transection or palsy that may cause de-innervation of muscles planned for implantation
* allergy to implanted materials
* existing active implant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Grip Accuracy | The measure will be carried out 11 times during the study, at Baseline with the subject's own device for comparison, and at 10 study visits with the investigational device conducted over approximately 6 months.
  Self-drafted assessment of accuracy in prosthesis movements. The purpose of this measure is to quantify subjects' ability to use the investigational device to control specific prosthetic movements. When performing the Accuracy Test, the subject attempts to execute a series of specified wrist and hand movements using the investigational device. An objective rater scores each movement on a 0-3 scale with 0 = no movement observed and and 3 = movement observed (with no unintended movements). A score is given for each movement and a combined score is derived from the complete set of movements.
  Administered as a repeated measure, the Grip Accuracy test assesses Change over time (training effect).

CONTACTS AND LOCATIONS:
Overall Officials: Aidan Roche, MD, Principal Investigator — NHS; University of Edinburgh
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No